CLINICAL TRIAL: NCT02907294
Title: Randomized, Double Blind, Placebo Controlled, Parallel Groups Study to Assess the Safety, Tolerability and Pharmacokinetic Profile of PBF-999 (160 mg and 320 mg) "After Multiple Oral Doses" in Healthy Volunteers
Brief Title: Study to Assess the Safety, Tolerability and Pharmacokinetic Profile of PBF-999 "After Multiple Oral Doses" in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: change in the therapeutic indication
Sponsor: Palobiofarma SL (Industry)
Collaborators: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIBSP-PBF-2015-82; 2015-004748-20 (EudraCT Number)
Record Dates: First submitted 2016-03-08; First posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Huntington Disease
Keywords: PDE10 inhibitor; phosphodiesterase 10 inhibitor; Huntington's disease; psychiatric disorders
MeSH Terms: conditions — Huntington Disease; Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PBF-999 (Experimental)
  Interventions: Drug: PBF-999 / 160 mg; Drug: PBF-999 / 320 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PBF-999 / 160 mg — 2 capsule 80 mg x 8 days
  Arms: PBF-999
Drug: PBF-999 / 320 mg — 4 capsule 80 mg x 8 days
  Arms: PBF-999
Drug: Placebo — 2 capsules of placebo x 8 days 4 capsules of placebo x 8 days
  Arms: Placebo

SUMMARY:
To assess the safety and tolerability of five doses of PBF-999 (160 mg and 320mg) after repeated (8 days) single daily oral dose administration in young male and female healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or females subjects, 18-45 years (inclusive) of age at the time of enrollment.
* Females must be of non-childbearing potential (i.e., surgically sterile) or have to use contraceptive measures (non-hormonal) such as condom, diaphragm or cervical/vault cap with spermicide until 28 days post-administration. Males should agree to abstain from sexual intercourse with a female partner or agree to use a condom with spermicide, in addition to having their female partner use some contraceptive measures until 28 days post-administration.
* Clinically acceptable blood pressure and pulse rate in supine and standing position. Blood pressure and pulse will be measured after a minimum of 3 minutes of resting.
* Body weight within normal range (Quetelet's index between 19 and 26) expressed as weight (kg) / height (m2).
* Able to understand the nature of the study and comply with all their requirements.
* Free acceptance to participate in the study by obtains signed informed consent form approved by the Ethics Committee of the Hospital (CEIC).

Exclusion Criteria:

* History of serious adverse reactions or hypersensitivity to any drug.
* Presence or history of allergies requiring acute or chronic treatment (except seasonal allergic rhinitis).
* Background or clinical evidence of chronic diseases.
* Acute illness two weeks before drug administration.
* Having undergone major surgery during the previous 6 months.
* Smokers (refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc., for 6 months prior to the administration of the study medication
* History of alcohol dependence or drug abuse in the last 5 years or daily consumption of alcohol > 40 g for men or 24 gr/day for women or high consumption of stimulating beverages (> 5 coffees, teas or coca cola drinks/ day)
* Abnormal physical findings of clinical significance at the screening examination or baseline which would interfere with the objectives of the study.
* Need of any prescription medication within 14 days prior to the administration of the drug and non prescription medication or herbal medicines within 7 days prior to the administration of the drug.
* Participation in other clinical trials during the previous 90 days in which an investigational drug or a commercially available drug was tested.
* Having donated blood during 4 weeks period before inclusion in the study.
* Existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the drug, i.e. impaired renal or hepatic function, diabetes mellitus, cardiovascular abnormalities, chronic symptoms of pronounced constipation or diarrhea or conditions associated with total or partial obstruction of the urinary tract.
* 12 lead ECG obtained at screening with PR ≥ 220 msec, QRS ≥120 msec and QTc ≥ 440 msec, bradychardia (<50 bpm) or clinically significant minor ST wave changes or any other abnormal changes on the screening ECG that would interfere with measurement of the QT interval.
* Symptoms of a significant somatic or mental illness in the four week period preceding drug administration.
* History of hepatitis HBV and / or HCV and / or positive serology results which indicate the presence of hepatitis B surface antigen and / or detectable HCV ribonucleic acid (RNA).
* Positive results from the HIV serology.
* Females with positive results from the pregnancy test or breast-feeding
* Clinically significant abnormal laboratory values (as determined by the Principal Investigator) at the screening evaluation.
* Positive results of the drugs at screening period or the day before starting treatment period. A minimum list of drugs that will be screened for include Amphetamines, Cocaine, Ethanol, Opiates, Cannabinoids and Benzodiazepines (positive results may be repeated at the discretion of the Principal Investigator).
* Known hypersensitivity to the study drug or the composition of the galenical form
* History of psychiatric diseases or epileptic seizures

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | from day 0 to day 15
  Vital Signs, ECG recordings, laboratory safety test and physical examination will be performed

SECONDARY OUTCOMES:
AUC | from day 1 to 8
  Day 1: baseline [pre-dose], [+10 min], [+20 min], [+40min], [+60min], [+ 1.5h], [+2 h], [+ 2.5 h], [+ 3 h], [+ 4h], [+8h], [+ 12h] and [+16h] post-medication;
  * Days 2 to 7: baseline [daily pre-dose] which corresponds at +24h of previous dose;
  * Day 8: baseline [daily pre-dose], [+10 min], [+20 min], [+40min], [+60min], [+1.5h], [+2 h], [+ 2.5 h], [+ 3 h], [+ 4h], [+8h], [+ 12h] and [+16h] and [+ 24h] post-daily medication (D9).
Cmax | from day 1 to 8
  Day 1: baseline [pre-dose], [+10 min], [+20 min], [+40min], [+60min], [+ 1.5h], [+2 h], [+ 2.5 h], [+ 3 h], [+ 4h], [+8h], [+ 12h] and [+16h] post-medication;

OTHER OUTCOMES:
Leeds Sleep Evaluation Questionnaire | from day 1 to 8
-Analogic visual scales (VAS/100) | from day 1 to 8
  ten scales will be used, Liking (only at +24 of the last drug administration), high, good effects, bad effects, sedation, nervous, euphoria, absent, vigouros and aphatetic.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Martinez, MD, Principal Investigator — CIM-Sant Pau
Locations (1):
- CIM-Sant Pau, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: phase 1 unit website — http://www.iibsantpau.cat/